CLINICAL TRIAL: NCT02851186
Title: Combined Electroacupuncture and Auricular Acupuncture for Postoperative Pain After Abdominal Surgery for Gynecological Diseases: A Randomized Sham-controlled Trial
Brief Title: Acupuncture for Postoperative Pain After Abdominal Surgery for Gynecological Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UW 15-459
Record Dates: First submitted 2016-07-19; First posted 2016-08-01 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroacupuncture (EA) and Auricular Acupuncture (AA) (Experimental): Subjects in the treatment group will receive EA combined with AA two hours before operation, immediately post-operation and once a day for the subsequent 5 days.
  Interventions: Device: Acupuncture
- Sham acupuncture (Sham Comparator): Subjects in the control group will receive non-invasive sham procedure in the same schedule as the treatment group.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture
  Arms: Electroacupuncture (EA) and Auricular Acupuncture (AA)
Device: Sham acupuncture
  Arms: Sham acupuncture

SUMMARY:
Objectives:

To examine the efficacy and safety of electroacupuncture (EA) combined with auricular acupuncture (AA) in reducing post-operative pain in patients following abdominal surgery for gynecological diseases.

Hypothesis:

Acupuncture is effective and safe to reduce postoperative pain during the first 5 days following surgery as compared to a sham control.

Design and strategy:

This is a randomized, placebo-controlled, subject- and assessor-blind trial. Seventy-two subjects will be recruited and randomized (in 1:1 ratio) to receive either acupuncture treatment or sham control. Subjects in both groups will undergo standard operation procedure and receive post-operative analgesics based on usual care.

Study instrument:

A 10-point pain Numerical Rating Scale (NRS) will be employed as a primary outcome assessment.

Intervention:

Subjects in the treatment group will receive EA combined with AA within two hours before operation, post-operation upon arrival to the ward and once a day for the subsequent 5 days. Subjects in the control group will receive non-invasive sham procedure in the same schedule.

Main outcome measures:

Primary outcome: NRS pain scores will be measured upon recovery, hourly at 6 hours after surgery, then 4-hourly until day 2, 6-hourly until day 3 and once daily until discharge.

Secondary outcome:

Morphine consumption, post-operative syndromes, quality of recovery questionnaire, SF-6D, EQ-5D-5L and adverse events will be documented and compared between groups.

Data analysis: Pain intensity during the first 5 days will be calculated by Area Under the Curve (AUC) of NRS pain scores. AUC between the two groups will be compared by Student's T-test.

Expected outcome: AUC of the acupuncture group is expected to be significantly lower than sham acupuncture group.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I to III
* Eligible for laparotomy with midline incision for gynaecological neoplasm including ovarian mass, uterine mass and cervical lesions
* Age 18 years or above
* Ability to understand the nature of the study and willing to give informed consent
* Capable of providing responses during outcome measurement

Exclusion Criteria:

* Having chronic pain and using any medication in addition to the anaesthetic and analgesia prescribed prior to surgery that would be expected to affect the dosage of postoperative analgesia
* History of or current alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120µmol/L
* Impaired hepatic function, defined as preoperative serum albumin level below 30g/L
* Impaired or retarded mental state and not able to sign the consent
* Not self-ambulatory before operation
* Difficulties in using patient-controlled analgesia
* BMI > 35kg/m2
* Infection observed at the acupoint sites
* History of acupuncture experience in the previous 12 months
* History or clinical evidence of valvular heart defects, heart failure, atrial fibrillation or bleeding disorders or are fitted with cardiac pacemaker or taking anticoagulant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve of Pain intensity by numerical rating scale (NRS) from baseline to day 5 | 5 days

SECONDARY OUTCOMES:
Pain intensity by numerical rating scale (NRS) at rest | Through study completion, an average of 7 days
Pain intensity by numerical rating scale (NRS) while coughing | Through study completion, an average of 7 days
Cumulative morphine consumption | Through study completion, an average of 7 days
Dose of rescues analgesic (IM morphine) use | Through study completion, an average of 7 days
Frequency of rescues analgesic (IM morphine) use | Through study completion, an average of 7 days
Time of recovery from postoperative syndrome | Through study completion, an average of 7 days
Quality of recovery (QoR-9) | Through study completion, an average of 7 days
SF-6D | Through study completion, an average of 7 days
EQ-5D-5L | Through study completion, an average of 7 days

OTHER OUTCOMES:
Number of patients withdraw | Through study completion, an average of 7 days
Reasons of withdrawal | Through study completion, an average of 7 days
Number of subjects with adverse events | Through study completion, an average of 7 days
Treatment Credibility by the Credibility of Treatment Rating Scale (CTRS) | Through study completion, an average of 7 days
Blinding Success Assessment by questionnaire | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Lixing LAO, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Kwong Wah Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong

REFERENCES:
- [Derived] Lam WL, Yeung WF, Wong MK, Cheung CW, Chan KKL, Ngan HYS, Wong CKH, Chen HY, Lao L. Combined electroacupuncture and auricular acupuncture for postoperative pain after abdominal surgery for gynecological diseases: study protocol for a randomized controlled trial. Trials. 2018 Jan 4;19(1):8. doi: 10.1186/s13063-017-2359-8. PMID 29301556